CLINICAL TRIAL: NCT03949270
Title: BETA-Text: Evaluating the Efficacy of a Novel, Interactive, Bidirectional Text-messaging Application to Increase Persistence to Adjuvant Endocrine Therapy for Stage I-III Hormone Receptor Positive Breast Cancer
Brief Title: Text Messaging in Patients on Adjuvant Endocrine Therapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000024495
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Adherence, Medication; Side Effect
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients in the usual care arm will not receive any text messages.
- BETA-Text Intervention (Experimental): Patients in the text messaging arm will receive daily, weekly, and monthly text messages.
  Interventions: Behavioral: BETA-Text text messaging intervention

INTERVENTIONS:
Behavioral: BETA-Text text messaging intervention — Patients in the text messaging arm will receive daily, weekly, and monthly text messages. The daily message asks whether or not the patient has taken their breast cancer medication. The weekly message asks about any side effects and their severity. The monthly text message asks about any barriers that the patient might be experiencing. Concerning responses to any of the text messages will prompt contact from the office of the treating physician.
  Arms: BETA-Text Intervention

SUMMARY:
1. The primary objective is to compare rates of persistence (continuation) of any endocrine therapy (ET) between patients assigned to standard of care follow-up (control arm) versus standard of care plus a bi-directional text messaging intervention (intervention arm)
2. The secondary objectives are:

   (i) To assess time to permanent discontinuation of ET (switching from an aromatase inhibitor to another ET is permitted). The investigators will also account for treatment breaks.

   (ii) To assess QOL at baseline, and at 6 and 12 months after initiation of ET (FACT-ES1, Brief Pain Inventory2, Overall Treatment Burden3,4, individual symptom LASA scales4) and compare between arms (iii) To assess adherence self-efficacy (SEAMS5 tool, Voils Extent of Non-Adherence Scale6), financial burden (COST tool7,8), beliefs about medications (modified BMQ tool9,10), and perceived ability to communicate with one's physician (PEPPI11 tool) and compare between arms (iv) To compare the time to endocrine therapy discontinuation in both the intervention and control arms (v) To characterize factors (including clinicopathologic features, socioeconomic status, and comorbidities) associated with non-adherence in both the intervention arm and the control arm, which may enable us to identify women who are at particularly high risk of non-adherence.

   (vi) To assess adherence to medication as reported through the BETA-Text intervention (vii) To collect the time to onset and trend of severity of side effects in women assigned to the text messaging intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed stage I-III, estrogen and/or progesterone receptor positive, as defined by ASCO-CAP guidelines, invasive breast cancer for whom adjuvant hormonal therapy is indicated following standard NCCN practice guidelines.42
2. Patients must initiate an aromatase inhibitor (AI), with the choice of AI (letrozole, anastrozole, or exemestane) left to the discretion of the treating provider (have just started or plan to start within 4 weeks)
3. Patients with synchronous bilateral breast cancers are eligible if both tumors are hormone receptor positive.
4. Patient must be able to provide informed consent and agree to:

   1. Complete questionnaires according to the pre-specified study design
   2. Own or have access to a personal cell phone, agree to send and receive text messages (including any costs), and share their personal cell phone number to receive text messages.
   3. Be able to read/speak English
   4. To allow research staff to contact their pharmacies to determine prescription refill dates.

Exclusion Criteria:

1. Patients with history of prior stage I-III breast cancer in the same or contralateral breast are not eligible (because exposure to prior endocrine therapy may confound results)
2. Patients with metastatic breast cancer.
3. Patients with ductal carcinoma in situ (DCIS) or other pre-malignant lesions of the breast receiving endocrine therapy as chemoprevention.
4. Prior treatment with an aromatase inhibitor, regardless of indication.
5. Prior tamoxifen for the current cancer (prior tamoxifen for DCIS or a different cancer is permitted).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Persistence to endocrine therapy at one year | 1 year

SECONDARY OUTCOMES:
Time to discontinuation of endocrine therapy | 1 year
Patient-reported Quality of life | 1 year
  FACT-ES (45 items). The survey assesses items on a 0-4 scale, where 0 is lack of a symptom and 4 is high degree of a symptom. There are 5 domains: physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and additional concerns/symptoms (14 items).
Pain (worst, least, current, average, and interference of pain) | 1 year
  Brief Pain Inventory (15 items), which measures worst pain, average pain, least pain, current pain, and pain interference on a 0-10 scale, where higher numbers indicate higher levels of pain.
Treatment Burden | 1 year
  Overall Treatment Burden (1 item), which assess the overall burden of treatment on a 0-100 visual analog scale. Higher numbers are indicative of higher treatment burden.
Self-Reported Adherence | 1 year
  Voils Extent of Non-Adherence Tool (3 items); items are scored 1-5; however, responses are dichotomized into either "adherent" (1) or "non-adherent" (2-5). A respondent must answer "1" for all three questions in order to be classified as "adherent"
Reasons for Non-Adherence | 1 year
  Voils Reasons for Non-Adherence Tool (24 items). Each item is measured on a scale of 1-5, with higher scores indicating more agreement with the particular item.
Adherence self-efficacy | 1 year
  SEAMS Questionnaire (13 items); items are scored 1-3 (range 13-39); the higher the score, the higher the self-efficacy of taking medication
Financial burden | 1 year
  COST tool (11 items); items are scored 0-4, some items are reverse scored; the lower the score, the worse the financial toxicity.
Beliefs about medication | 1 year
  BMQ tool (18 items); assessing patients' beliefs about the necessity of prescribed medication for controlling their illness and their concerns about the potential adverse consequences of taking it; higher scores indicate stronger beliefs in the concepts represented by the scale. There are an additional 8 questions which similarly address Overuse and Harm.
Communication with one's physician | 1 year
  PEPPI instrument (5 items); range of scores 5-25, where high scores indicate patient-reported better patient-physician communication and interaction
Time to onset and trend of severity of side effects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mougalian, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mougalian SS, Epstein LN, Jhaveri AP, Han G, Abu-Khalaf M, Hofstatter EW, DiGiovanna MP, Silber ALM, Adelson K, Pusztai L, Gross CP. Bidirectional Text Messaging to Monitor Endocrine Therapy Adherence and Patient-Reported Outcomes in Breast Cancer. JCO Clin Cancer Inform. 2017 Nov;1:1-10. doi: 10.1200/CCI.17.00015. PMID 30657377